CLINICAL TRIAL: NCT04325646
Title: Sero-epidemiological Study of the SARS-CoV-2 Virus in France: Constitution of a Collection of Human Biological Samples
Brief Title: Sero-epidemiological Study of the SARS-CoV-2 Virus Responsible for COVID-19 in France
Acronym: CORSER
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-007
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: SARS (Severe Acute Respiratory Syndrome); COVID-19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, nasal swab, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- CORSER-1a: Subjects who had been to China in the weeks before the outbreak began
  Interventions: Other: Human Biological samples
- CORSER-1b: Subject who had a clinical profile compatible with an SARS-CoV-2 infection between August 1, 2019 and February 29, 2020
  Interventions: Other: Human Biological samples
- CORSER-2a: Subjects with suspected CoV-2-SARS infection with negative results from RT-PCR testing of respiratory specimens
  Interventions: Other: Human Biological samples
- CORSER-2b: Contacts or co-exposures of confirmed CoV-2-SARS infection cases, or who have worked or stayed in a hospital where confirmed CoV-2-SARS infection has been managed
  Interventions: Other: Human Biological samples
- CORSER-2c: Subjects who have been exposed to a risk of infection with SARS-CoV-2 in a geographical area of SARS-CoV-2 circulation.
  * study among pupils, their parents and siblings, as well as teachers and non-teaching staff of a high-school located in Oise
  * study among pupils from 5 to 12 and their parents in elementary schools located in Oise
  * study among choir members
  Interventions: Other: Human Biological samples
- CORSER-2d: Staff of health care institutions
  Interventions: Other: Human Biological samples
- CORSER-2e: Subjects in care, hospitalized or residing in health care facilities
  Interventions: Other: Human Biological samples
- CORSER-3: Subjects returning from a humanitarian mission that started before 31/01/2020
  Interventions: Other: Human Biological samples
- CORSER-2f: Subjects with two symptomatic episodes of SARS-CoV-2 infection
  Interventions: Other: Human Biological samples
- CORSER-4: Subjects being vaccinated against COVID-19
  Interventions: Other: Human Biological samples
- CORSER-5: Subjects with acute SARS-CoV-2 infection and uninfected controls
  Interventions: Other: Human Biological samples

INTERVENTIONS:
Other: Human Biological samples — Blood samples for serological tests
  Groups: CORSER-1a; CORSER-1b; CORSER-2a; CORSER-2b; CORSER-2c; CORSER-2d; CORSER-2e; CORSER-3
Other: Human Biological samples — Blood samples, saliva, nasopharyngeal swab for serological tests
  Groups: CORSER-2f; CORSER-4; CORSER-5

SUMMARY:
On January 2020, the discovery of a new coronavirus (SARS-CoV-2) was officially announced by the Chinese health authorities and the World Health Organization (WHO). Its complete genome was sequenced by the laboratory of respiratory infection viruses at the Institut Pasteur on 29 January 2020 in France. This will allow the identification of antigenic structures involved in the immune response and the development of serological diagnostic tests.

Many questions are being asked about this new virus and the infection it causes, including questions about the percentage of asymptomatic and pauci-symptomatic forms. Serological studies can provide answers to these questions. There is no serological test for SARS-COV-2 yet, but the laboratory of respiratory infection viruses at the Institut Pasteur is working on its development.

This study proposes to carry out a collection of samples taken from subjects who travelled to China before the epidemic outbreak or suspected of being infected with SARS-CoV-2.

As soon as it is available, serology will be performed on the collected samples.

DETAILED DESCRIPTION:
On January 2020, the discovery of a new coronavirus (SARS-CoV-2) was officially announced by the Chinese health authorities and the World Health Organization (WHO). This new virus is presented as the causative agent of pneumonias. Its complete genome was sequenced by the laboratory of respiratory infection viruses at the Institut Pasteur on 29 January 2020 in France. This will allow the identification of antigenic structures involved in the immune response and the development of serological diagnostic tests.

Many questions are being asked about this new virus and the infection it causes, including questions about the transition from animal to human occur, the beginning of viral circulation in humans, the period of contagiousness, the percentage of asymptomatic and pauci-symptomatic forms. Serological studies can provide answers to these questions. There is no serological test for SARS-COV-2 yet, but the laboratory of respiratory infection viruses at the Institut Pasteur is working on its development.

This study proposes to carry out a collection of samples taken from subjects who travelled to China before the epidemic outbreak or suspected of being infected with SARS-CoV-2.

As soon as it is available, serology will be performed on the collected samples.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with or benefiting from a Social Security system
* State of health compatible with a blood sample as defined in the protocol

Exclusion Criteria:

* Person benefiting from a legal protection measure or unable to express informed consent to participation
* Have had an infectious episode and/or respiratory signs in the 14 days prior to the scheduled visit (CORSER 1 and 2a, 2b)
* Have been in contact with a confirmed case of SARS-CoV-2 infection within 14 days prior to the date of the visit.(CORSER 1 and 2a, 2b)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults (≥ 18 years old) at the time of collection (including minors for group 2c)
  CORSER-1 : subjects who were in China between 08/2019 and 01/2020 and who have not been diagnosed with an SARS-CoV-2 infection;
  CORSER-2 :
  Sub-group 2a: suspected SARS-CoV-2 infection with a negative result of RT-PCR virus test on respiratory sample.
  Sub-group 2b: contact or co-exposure with confirmed cases of SARS-CoV-2-infection.
  Subgroup 2c: exposed to a risk of infection with SARS-CoV-2 in a geographic area of SARS-CoV-2 circulation.
  Subgroup 2d : Staff of health care institutions
  Subgroup 2e : hospitalized or residing in health care facilities
  Subgroup 2f : Subjects with two symptomatic episodes of SARS-CoV-2- infection
  CORSER 3 : returning from a humanitarian mission that started before the epidemic circulation of the virus in France
  CORSER 4 : being vaccinated against COVID-19
  CORSER 5 : with acute SARS-CoV-2 infection and controls
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Presence of specific anti-SARS-CoV-2 antibodies in the different study groups. | One year
  Description of the serological status of individuals by different detection tests

SECONDARY OUTCOMES:
Percentage of asymptomatic forms in individuals with anti-SARS-CoV-2 antibodies | One year
  Proportion of asymptomatic subjects into seropositive population

CONTACTS AND LOCATIONS:
Overall Officials: Bruno HOEN, Pr, Principal Investigator — Institut Pasteur
Locations (21):
- France (21):
  - CHU Amiens-Picardie, Amiens
  - EHPAD Villa Concorde, Asnières-sur-Seine
  - CHU François Mitterand, Dijon
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - CHU Limoges, Limoges
  - Hôpital de la Croix Rousse, Lyon
  - EHPAD Les Etangs, Mennecy
  - CHRU de Nancy, Nancy
  - Hôpitaux de Brabois, Nancy
  - CHR Orléans, Orléans
  - Institut Mutualiste, Paris
  - Centre Médical de l'Institut Pasteur, Paris
  - Institut Pasteur, Paris
  - EHPAD Villa Lecourbe, Paris
  - Hôpital la Pitié Salpetrière, Paris
  - CHU Poitiers, Poitiers
  - Hôpital Pontchaillou, Rennes
  - CHU Saint-Etienne, Saint-Etienne
  - CHRU de Strasbourg, Strasbourg
  - CH de Tourcoing, Tourcoing
  - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia L, Woudenberg T, Rosado J, Dyer AH, Donnadieu F, Planas D, Bruel T, Schwartz O, Prazuck T, Velay A, Fafi-Kremer S, Batten I, Reddy C, Connolly E, McElheron M, Kennelly SP, Bourke NM, White MT, Pelleau S. Kinetics of the SARS-CoV-2 Antibody Avidity Response Following Infection and Vaccination. Viruses. 2022 Jul 8;14(7):1491. doi: 10.3390/v14071491. PMID 35891471
- [Derived] Benetos A, Lai TP, Toupance S, Labat C, Verhulst S, Gautier S, Ungeheuer MN, Perret-Guillaume C, Levy D, Susser E, Aviv A. The Nexus Between Telomere Length and Lymphocyte Count in Seniors Hospitalized With COVID-19. J Gerontol A Biol Sci Med Sci. 2021 Jul 13;76(8):e97-e101. doi: 10.1093/gerona/glab026. PMID 33528568